CLINICAL TRIAL: NCT01379313
Title: The Effect of Different I:E Ratio on Gas Exchange of Patients Undergoing Gynecologic Laparoscopic Surgery With Trendelenburg Position
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Tae Soo Hahm, Professor, Samsung Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 2011-04-007
Record Dates: First submitted 2011-06-21; First posted 2011-06-23 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Uterine Myoma; Ovarian Cyst; Laparoscopic Gynecologic Surgery
Keywords: laparoscopic gynecologic surgery; gas exchange; inspiratory time; expiratory time; I:E ratio
MeSH Terms: conditions — Myofibroma; Ovarian Cysts | interventions — Buspirone; Population Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1:2 group (Active Comparator): conventional I:E ratio group, inspiratory time : expiratory time = 1:1
  Interventions: Procedure: conventional I:E ratio
- 1:1 group (Experimental): 1:1 I:E ratio group, inspiratory time : expiratory time = 1:1
  Interventions: Procedure: 1:1 ratio
- 2:1 group (Experimental): inverse ratio group, inspiratory time : expiratory time = 2:1
  Interventions: Procedure: 2:1 group
- 1:2 PEEP group (Active Comparator): I:E ratio of 1:2 with external PEEP of 5 cm H2O
  Interventions: Procedure: conventional I:E ratio; Procedure: external PEEP

INTERVENTIONS:
Procedure: conventional I:E ratio — conventional I:E ratio of 1:2 is applied.
  Arms: 1:2 PEEP group; 1:2 group
Procedure: 1:1 ratio — I:E ratio of 1:1 is applied.
  Arms: 1:1 group
Procedure: 2:1 group — Inverse I:E ratio of 2:1 is applied.
  Arms: 2:1 group
Procedure: external PEEP — external positive end-expiratory pressure of 5 cmH2O is applied.
  Arms: 1:2 PEEP group

SUMMARY:
In patients undergoing gynecologic laparoscopic surgery with trendelenburg position, the disturbance of pulmonary gas exchange frequently occurs due to high intra-abdominal pressure. The investigators tried to evaluate the effect of various inspiratory to expiratory ratio on pulmonary gas exchange by randomized controlled trial.

DETAILED DESCRIPTION:
In patients undergoing gynecologic laparoscopic surgery with trendelenburg position, the disturbance of pulmonary gas exchange frequently occurs due to high intra-abdominal pressure. During the laparoscopic surgery with abdominal gas insufflation, gas exchange disturbance such as CO2 retention, hypoxemia occurs in addition to high plateau airway pressure. The usual strategy against these kinds of problem is pressure-controlled ventilation. However, the gas exchange problem especially CO2 retention can not be solved in some cases. The inverse-ratio ventilation (IRV), which prolongs the inspiratory time greater than expiratory time, can be applied for adult respiratory distress syndrome. The efficacy of IRV is to improve gas-exchange status by increasing mean airway pressure and alveolar recruitment. There have been several clinical investigations which applied IRV during general anesthesia. However, there have been debates about the effect of IRV during general anesthesia. Therefore, we tried to apply the IRV for subjects undergoing laparoscopic surgery, and evaluate the effect of different I:E ratio on the pulmonary gas exchange and respiratory mechanics.

ELIGIBILITY:
Inclusion Criteria:

* patients undergoing elective gynecologic laparoscopic surgery
* the duration of pneumoperitoneum during laparoscopic surgery is more than 40 minutes

Exclusion Criteria:

* ASA (American society of anesthesiologists) classification of the subjects more than III.
* Age under 20, or more than 65 years.
* Past history of pneumothorax, COPD, asthma.
* Patients with ischemic heart disease, valvular heart disease.

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2011-06; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
arterial CO2 partial pressure | 10 minutes after induction of general anesthesia
  arteial CO2 partial pressure
arterial CO2 partial pressure | 30 minutes after start of pneumoperitoneum
  arteial CO2 partial pressure
arterial CO2 partial pressure | 60 minutes after start of pneumoperitoneum
  arteial CO2 partial pressure

SECONDARY OUTCOMES:
arterial O2 partial pressure | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  arterial O2 partial pressure
Mean airway pressure | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  Mean airway pressure
tidal volume (setting) | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  tidal volume (setting)
hemodynamic parameters | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  systolic/ diastolic blood pressure, heart rate, mean blood pressure
end-tidal CO2 partial pressure | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  end-tidal CO2 partial pressure
respiratory compliance | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  Dynamic compliance, Static compliance
Dead space | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  physiologic dead space / tidal volume (VD/VT)
work of breathing | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  work of breathing
peak inspiratory pressure | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  peak inspiratory pressure
plateau pressure | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  plateau pressure
positive end-expiratory pressure | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  positive end-expiratory pressure
tidal volume (exhaled) | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  tidal volume (exhaled)
minute ventilation | 10 min after induction, 30 and 60 min after start of pneumoperitoneum
  minute ventilation

CONTACTS AND LOCATIONS:
Overall Officials: Tae Soo Hahm, M.D.,Ph.D., Study Director — Samsung Medical Center; Won Ho Kim, M.D., Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Seoul Hospital, Samsung Medical Center, Seoul, South Korea